CLINICAL TRIAL: NCT04433884
Title: Evaluation of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation Using Conventional Laryngoscope Versus C-MAC Video Laryngoscope in Patients Undergoing Elective Coronary Artery Bypass Grafting (CABG) Surgery - A Randomized Control Trial.
Brief Title: Evaluation of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation Using Conventional Laryngoscope Versus C-MAC Video Laryngoscope in Patients Undergoing Elective Coronary Artery Bypass Grafting (CABG) Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sehrish khan, Resident, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-3278-9046
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Intubation Complication

STUDY DESIGN:
Who Masked: Participant
Masking Description: Computer generated randomization using envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional MAC Laryngoscope (Experimental): Patients in this group will undergo intubation using conventional macintosh laryngoscope
  Interventions: Device: Endotracheal intubation using a laryngoscope
- C-MAC Video laryngoscope (Experimental): Patients in this group will undergo intubation using video C-Mac laryngoscope
  Interventions: Device: Endotracheal intubation using a laryngoscope

INTERVENTIONS:
Device: Endotracheal intubation using a laryngoscope — Patients will undergo intubation using 2 different types of laryngoscopes and their hemodynamic response would be recorded

SUMMARY:
This study is being done to compare hemodynamic response upon endotracheal intubation using either conventional laryngoscopy with Macintosh blade versus C-Mac video laryngoscope in patients undergoing elective coronary artery bypass grafting without anticipated difficult airway.

DETAILED DESCRIPTION:
Patients will be premeditated with 7.5mg oral midazolam approximately 45-60 minutes prior to anesthesia. The standard monitoring of Electrocardiography for ST analysis and SPO2 will be monitored continuously. Capnography, tidal volume and airway pressure will also be monitored during anesthesia. Arterial line for invasive Blood Pressure monitoring, wide bore IV cannula will be placed before induction of anesthesia. Anesthesia technique will be standardized in both groups. After pre-oxygenation, anesthesia co-induction will be done with midazolam 0.02-0.05 mg/kg, propofol 0.5-1mg/kg and fentanyl 5mcg/kg. Cis-atracurium 0.15mg/kg will be used as muscle relaxant. Patient will be ventilated manually by using isoflurane (1% end tidal) in oxygen using facemask. ETT will be placed orally via direct laryngoscopy by MC and C-MAC blade 3 or 4 when a Train of Four would not be achieved. All intubation will be performed by senior experienced anesthetist having experience of at least 20 intubations using video laryngoscope.

After induction a central venous catheter will be placed for central venous pressure monitoring and a thermo dilution Swan Ganz catheter will be inserted if indicated.

Tracheal intubation will be performed using the standard Macintosh laryngoscope(MC) or C- MAC video laryngoscope (VL) (Karl Storz, Tuttlingen, Germany).

Hemodynamic changes, laryngoscopic view, the number of attempts, the time required for laryngoscopy and tracheal intubation, changes in rhythm, and intraoperative and post operative complications will be recorded. Heart rate (HR), systolic arterial pressure (SAP), diastolic arterial pressure (DAP) and mean arterial pressure (MAP) along with peripheral oxygen saturation (SpO2), will be recorded before (T1) and after induction (T2), 1 minute after intubation (T3), 5 min (T4) and 10 min (T5)post intubation. End tidal carbon dioxide (EtCO2) will be recorded immediately after induction (T2), immediately after intubation 1 minute (T3), 5 min (T4) and 10 min (T5) post intubation. Measurements obtained after induction of anesthesia when the hemodynamics will be stable (post induction) will be considered as baseline measurements in the study.

Duration of laryngoscopy (DOL) is defined as the time from oral placement of the laryngoscope blade to obtaining the best glottic view. For the evaluation of glottic view during laryngoscopy, modified Cormack and Lehane Scoring System (m CL) and percentage of the glottis opening (POGO) score will be used. Duration of intubation (DOI) is defined as the time interval between oral placement of the ET to the attainment of tracing of 3 EtCO2 waveforms after intubation and initiation of mechanical ventilation. An attempt is defined as the time from introduction of laryngoscope into the oral cavity until its removal. Three attempts at intubation will be allowed for all groups. Failure to intubate will be defined as the inability to intubate after three attempts. An alternative technique will be used in cases of failure as per the discretion of anesthetist. In the case of multiple attempts, the duration of each attempt will be recorded. The duration of laryngoscopy and intubation (DOLI) is defined as the sum of all intubation attempts. The hemodynamic changes after intubation will be evaluated after successful intubation. After the study period, the anesthetic agents will be used as per the patient requirement. A number of unsuccessful attempts of intubation, complications encountered during intubation (bleeding, lacerations, dental injury, etc.,), and optimal laryngeal external manipulation (OLEM) during intubation will be recorded. The management of these complications will be done by primary anaesthesia team as per their feasibility and the costs of management of these complications will be covered under hospital insurance. Difficult intubation will be assessed by using Intubation Difficulty score (Table 1), Thyromental distance and Upper lip bite test.

Adverse effects of A number unsuccessful attempts of intubation, complications encountered during intubation (bleeding, lacerations, dental injury, etc.,), and optimal laryngeal external manipulation (OLEM) during intubation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65
* Elective Coronary Artery By Pass Grafting
* American Society Of Anesthesiologist III/IV
* Unanticipated difficult airway
* Mallampati I-II

Exclusion Criteria:

* Obese Body Mass Index > 35kg/m2
* Left Main Coronary Artery critical Disease
* Recent MI or unstable Angina
* Left heart failure/ Left ventricular ejection fraction<35%
* Upper lip bite test class III
* Thyromental distance <6.0 cm
* Emergency surgery
* Anticipated difficult airway
* Respiratory Diseases
* Bleeding diathesis
* Neurological deficit
* Limited nuchal Range of motion
* Gastro Esophageal Reflux Disease

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-06-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure (in millimeters of Hg) | Baseline before induction, 1 minutes after intubation, 5 minutes after intubation, 10 minutes after intubation
  Hemodynamic response
Changes in heart rate (beats per minute) | Baseline before induction, 1 minutes after intubation, 5 minutes after intubation, 10 minutes after intubation
  Hemodynamic response

SECONDARY OUTCOMES:
Arrhythmias | Baseline before induction, 1 minutes after intubation, 5 minutes after intubation, 10 minutes after intubation
  Presence of arrhythmias would be noted
Perioperative myocardial ischemia | Baseline before induction, 1 minutes after intubation, 5 minutes after intubation, 10 minutes after intubation
  Presence of myocardial ischemia would be noted by ST segment changes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Karachi, Sindh, Pakistan